CLINICAL TRIAL: NCT04193228
Title: Exploring Muscle Structure, Function and Gait Patterns in People With Distal Hereditary Motor Neuropathy: Natural History and the Effect of Rehabilitation Interventions
Brief Title: Muscle Structure, Function and Gait in dHMN
Acronym: GAIT-dHMN
Status: Completed | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Gita Ramdharry, Consultant Allied Health Professional, University College London Hospitals
Other Study IDs: pending
Record Dates: First submitted 2019-10-23; First posted 2019-12-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Distal Hereditary Motor Neuropathy, Type II; Distal Hereditary Motor Neuropathy, Type V; Distal Hereditary Motor Neuronopathy Type I; Distal Hereditary Motor Neuronopathy Type VI
MeSH Terms: conditions — Distal Hereditary Motor Neuropathy, Type II; Neuronopathy, Distal Hereditary Motor, Type V; Neuronopathy, Distal Hereditary Motor, Type I; Spinal muscular atrophy with respiratory distress 1 | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with distal hereditary motor neuropathy: This is a single arm, feasibility study
  Interventions: Device: Carbon Fibre Ankle Foot Orthosis; Behavioral: Exercise

INTERVENTIONS:
Device: Carbon Fibre Ankle Foot Orthosis — Off teh shelf carbon fibre ankle foot orthoses worn bilaterally
  Other Names: Ankle Foot Orthosis
Behavioral: Exercise — Ankle muscle strength training

SUMMARY:
Distal Hereditary Motor Neuropathy (dHMN) is a rare inherited neuromuscular disorder. It is characterised by distal weakness. The condition usually manifests in the second decade of life and progresses slowly. Though patients usually have a normal lifespan it is a disabling condition and most eventually need aids to walk. In order to improve walking quality in patient with dHMN, research is needed to understand the impairments that lead to altered gait patterns, and to develop interventions to correct walking gait conservatively.

In this proposed trial our goal is to explore the relationships between muscle structure, function and gait patterns for people with Distal Hereditary Motor Neuropathy. Over 12 months, muscle changes in dHMN are going to be observed in terms of structure and function using MRI, myometry and 3D motion analysis. In addition, the effect of a 16 weeks exercises program on muscle structure and function in dHMN is going to be measured by the same observational methods. To address walking gait directly in dHMN, gait patterns with and without wearing carbon fibre ankle foot orthoses (AFO)will be measured using 3D motion analysis.

DETAILED DESCRIPTION:
Objectives: The primary objective (objective 1) is to:

1. explore the natural history of muscle structure and function in Distal Hereditary Motor Neuropathy (dHMN) over one year.

   The secondary objectives are:
2. to ascertain relationships between intramuscular fat fraction (measured by MRI), muscle volume, isokinetic muscle strength (measured by dynamometry) and moments/power generation (measured by 3D gait analysis) (objective 2).
3. to explore the effect of bilateral carbon fibre ankle foot orthoses (AFO) on the kinetics and kinematics of gait of people with DHMN (measured by 3D gait analysis) (objective 3).
4. to explore the effect of resistance training of the ankle muscles in people with ankle muscle strength over grade 4 MRC scale on muscle structure, function, and gait patterns (objective 4).

Type of trial: A prospective cohort study in adult patients with dHMN with a single UK site.

Trial design and methods: This study (participants with dHMN and control participants) is proposed to take place over 3 years in one site in the UK (NHNN). Participants with dHMN aged over 18 for potential enrolment in the study will be identified through existing inherited neuropathy cohort clinics at NHNN and healthy control participants will be invited. If they show interest in participating, they will be given the relevant Patient Information Sheets and Informed Consent Forms.

Objective 1&2: dHMN participants will undergo the following measures: MRI scans of the legs, isokinetic strength and power measures of the lower limb using the HUMAC Norm dynamometer,3D motion analysis to capture kinetic and kinematic data of complete gait cycles. Clinical assessments will be undertaken to measure: gait speed and endurance, joint range of motion, foot posture, pain and sensory impairment. For direct comparison of gait deviations, twenty age and gender matched health controls will also be recruited to undergo the same measures. Scans, dynamometry and clinical measures will be repeated after one year to explore the natural history of the disease.

Objective 3: The dHMN participants recruited for objective 1 will undergo additional gait analysis: wearing just shoes (control condition), wearing their own prescribed orthoses (where appropriate), and wearing bilateral carbon fibre AFOs. The order of wearing or not wearing the AFOs will be randomised to account for learning and/or fatigue effects.

Objective 4: The participants from objective 1 will be invited to participate in the strength training study and will be screened to see if they meet the inclusion criteria. The primary criteria will be that at least one of the major muscle groups of the ankle, dorsiflexors or plantarflexors, will score over 4/5 on the MRC scale. There might be a need for recruiting more participants if less than 10 from objective 1 participants met the inclusion criteria. Up to 15 participants will be prescribed a home based, resistance training trial for 16 weeks, supervised by the PhD candidate through weekly phone calls and monthly monitoring through an app, and progression visits. Response to training will be analysed by: MRI scans, myometry, and 3D motion analysis.

Trial duration per participant: 16 months Estimated total trial duration: 36 months Planned trial sites: The National Hospital for Neurology and Neurosurgery (NHNN), UCLH NHS Foundation Trust.

Total number of participants planned: 20 participants with dHMN and 20 matching control participants will be recruited for objective 1. Participates with dHMN will be invited to participate for objective 2 and 3.

Main inclusion/exclusion criteria: The main disease to be investigated is dHMN. The key inclusion criteria are: adult patients aged 18 or above with clinically proven dHMN; patients who are able to complete calf and thigh myometry, able to walk for 10 minutes without walking aids, and have no contraindication to MRI scanning. For objective 4, at least one of the major muscle groups of the ankle, dorsiflexors or plantarflexors, will score over 4/5 on the MRC scale. The key exclusion criteria are: patients having undergone lower limbs surgery in the year prior to the trial enrolment or planned to have lower limb surgery in the 16 months of the study; bilateral arthrodesis; participants having another medical condition which precludes them having an MRI scan; patients with a known diagnosis of another neurological disease. Control participants must have no known neuromuscular disease, have no contraindication to MRI scanning, be able to complete calf and thigh myometry and 3D gait analysis.

ELIGIBILITY:
Inclusion criteria for participants with dHMN

1. Adult patients aged 18 or above.
2. Clinical and electrophysiological features of dHMN.
3. Participant is able to give informed consent and has signed the informed consent form.
4. Patients who are able to complete calf and thigh myometry and 3D gait analysis.
5. Patients who have no contraindication to MRI scanning.
6. Participant for objective 3, at least one of the major muscle groups of the ankle, dorsiflexors or plantarflexors, will score over 4/5 on the MRC scale.

Inclusion criteria for control participants

1. Adult aged 18 or above.
2. Participants who have no known neuromuscular disease.
3. Participant is able to give informed consent and has signed the informed consent form.
4. Participants who are able to complete calf and thigh myometry and 3D gait analysis.
5. Participants who have no contraindication to MRI scanning

Exclusion criteria for dHMN participants:

1. Known neuromuscular disorder other than dHMN.
2. Lower limbs surgery planned during the study period or performed within the preceding 12 months.
3. Bilateral arthrodesis.
4. The participant has a contraindication for MRI scan.
5. Females who are pregnant, planning pregnancy or breastfeeding.

Exclusion criteria for Control participants:

1. The participant has a contraindication for MRI.
2. Participants who cannot complete calf and thigh myometry and 3D gait analysis.
3. Participant has a history, signs or symptoms of a neuromuscular disorder.
4. Females who are pregnant, planning pregnancy or breastfeeding.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with clinically confirmed distal hereditary motor neuropathy
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Muscle fat fraction | 16 weeks
  Percentage fat fraction measured by the 3-point Dixon method

SECONDARY OUTCOMES:
3D gait analysis | 16 weeks
  Kinematic measures: pelvis, hip, knee and ankle angular displacement during one gait cycle Kinetic: plantar flexor moment (Nm) and power generation (W) at pre-swing
Isokinetic muscle function | 16 weeks
  Isokinetic torque for lower limb flexors and extensors (Nm)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Square centre for Neuromuscular Diseases, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on request